CLINICAL TRIAL: NCT04030884
Title: The Effect of Oral Honey and Water Up to Two Hours Before Surgery on Postoperative Nausea and Vomiting
Acronym: PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OYA GUMUSKAYA BRADLEY (Other)
Responsible Party: Sponsor-Investigator, OYA GUMUSKAYA BRADLEY, Assistant Professor, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 03/05/2017-166977
Record Dates: First submitted 2019-07-08; First posted 2019-07-24 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: postoperative nausea and vomiting; nursing; oral carbohydrate; honey
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Honey

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with two types of surgery compared, each consisting intervention and control groups.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants were blinded regarding which gastrointestinal complication was going to be evaluated after the surgery. Participants were informed that the intervention was for postoperative gastrointestinal comfort, without nausea and vomiting being mentioned in order to avoid psychological leading to PONV.
  The nurses who collected the data were blinded for the group information (intervention or control) though they were informed the days of participant allocation (each morning they were informed that the current operating list included participants) for the proper use of the data collection forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention Lap.Chol. (Experimental): Honey and water mixture was ingested up to two hours preoperatively by the participants who were going to have a laparoscopic cholecystectomy.
  Interventions: Dietary Supplement: Honey and water mixture
- Control Lap.Chol. (No Intervention): The participants received standard care for their laparoscopic cholecystectomy.
- Intervention Thyroidectomy (Experimental): Honey and water mixture was ingested up to two hours preoperatively by the participants who were going to have a thyroidectomy.
  Interventions: Dietary Supplement: Honey and water mixture
- Control Thyroidectomy (No Intervention): The participants received standard care for their thyroidectomy.

INTERVENTIONS:
Dietary Supplement: Honey and water mixture — 60 gr of organic Turkish BlackSea Region Chestnut Honey and 100 ml Spring water mixture both mixed in room temperature and ingested up to two hours before the surgery by participants who were "nill by mouth" from midnight prior to the operation day.
  Arms: Intervention Lap.Chol.; Intervention Thyroidectomy

SUMMARY:
Postoperative nausea and vomiting (PONV) remains current as a complication and moderate evidence is available regarding the impact of preoperative oral carbohydrate-fluid administration on PONV. Honey, a natural source of carbohydrates, has an antioxidative effect and protects the gastric mucosa.

Aim: To investigate the effect of oral honey and water for up to 2 hours preoperatively on PONV.

Methods: A total of 142 elective thyroidectomy (experiment:35; control:37) and laparoscopic cholecystectomy (experiment:33; control: 37) patients were included. The experiment group was administered a 60 grams honey and 100 ml water mixture up to 2 hours preoperatively. The patients were monitored postoperative 0-6 hours using Rhodes Index of Nausea-Vomiting-Retching (R-INVR) and visual analog scale (VAS) for PONV.

DETAILED DESCRIPTION:
The American Society of PeriAnesthesiology Nurses (ASPAN) describes postoperative nausea and vomiting (PONV) as nausea and vomiting within the first 24 hours after an operation and early PONV for the first six hours. PONV is a frequent complication of surgical stress, extended fasting period and anaesthetic agents and has reported in 30% to 45% of patients, up to 80% of the patients at risk groups; especially for people who has gastrointestinal or major surgical procedures. Overall, one third of all patients who undergone a surgical intervention are said to experience PONV.

PONV causes discomfort, which may increase anxiety, and can induce indirect or direct pain in the individual. This may lead to an increase in intra-abdominal pressure, central venous pressure, blood pressure and intracranial pressure, increased risk of cardiac rhythm disturbances, and it can lead up to other complications such as risk of aspiration, a stretching of the incision. Therefore, the study was planned to evaluate as many variables as possible that affect PONV with the use of honey as a source of carbohydrate for the carbohydrate solutions (CS). By doing so, supplying carbohydrate to patients with a daily source of natural nutrient with its additional benefits of gastric mucosal protection was expected to decrease PONV. Honey has been widely used for its medicinal purposes for centuries and is suggested for daily intake for gastric protection. It was proved as an effective wound care material and rodent studies have showed outstanding results on gastric mucosa and ulcer treatment.

Hypothesis:

H1. The risk of PONV decreases with honey and water consumption in immediate preoperative period.

H2. Blood sugar level (BGL) is regulated as the fasting period is shortened in patients who receive honey orally.

Intervention:

The experiment group received 60 g honey in a 190 ml food grade empty glass jars which were topped with 100 ml room temperature drinking water and mixed. For standardization of the honey content, Turkish Black Chestnut Honey were purchased from a registered producer. The honey then was sent to be tested for safety and quality analysis and has found to be within the acceptable quality limits of international standards. This information was shared with participants.

The experiment and the control group both were observed for the first 6 hours after surgery by the post anaesthesia care unit (PACU) and ward nurses who were blinded to the group information.

Data Collection A data collection form consisting of 23 questions and sub-items including participants' demographics and questioning the risk of nausea and vomiting was prepared according to the related literature.

Data collection form;

1. The demographic chapter comprises; age, gender, educational status, height, weight, body mass index, general health status, allergies
2. Planned surgical intervention and anaesthesia applications; surgery, type and the duration of anaesthesia, anaesthetic agents,
3. Nausea and vomiting risk assessment questions of Koivuranta scale; age, gender, smoking status, previous nausea vomiting experience, the duration of anaesthesia,
4. Post-operative period; complications, a two-hour postoperative pain visual analogue scale (VAS), blood sugar levels, drugs for nausea and vomiting,
5. VAS and Rhodes Index of Nausea, Vomiting and Retching (R-INVR) to examine PONV. The Index of Nausea Vomiting and Retching was developed by Rhodes and McDaniel and adaptation, validity and reliability in Turkish population of the scale was carried out by Tan and Genç (2010).

The Statistical Analysis:

The statistical analysis was performed using IBM SPSS 21.0 (IBM Corp. released 2012, Armonk, NewYork, USA). Descriptive statistics; mean, standard deviation, median, smallest-largest, frequency, percent. In the comparison of discrete variables; Pearson's chi-square and Fisher's exact test were used. The suitability of continuous variables to normal distribution was evaluated by Kolmogorov Smirnov test. Intergroup comparisons of continuous variables were performed by Kruskal Wallis, independent samples t test and Mann Whitney U test. Bonferroni corrected Mann Whitney U test was used in paired group comparisons (post hoc) when the results of Kruskal Wallis test were meaningful. Intra-group comparisons were performed with t test in dependent groups. Pearson and Spearman correlation tests were used to evaluate the linear relationship between the variables. A p value of <0.05 was accepted for statistical significance.

ELIGIBILITY:
Inclusion Criteria

* Individuals who volunteered to participate in the study
* Individuals who have the ability to make decisions
* Thyroidectomy operation
* Laparoscopic cholecystectomy (Lap. Chol.) operation
* Individuals who score 2/5 or more out of the Koivuranta PONV risk factors*

Exclusion Criteria

* Patients with diabetes,
* Nothing by mouth patients (for other reasons than surgery),
* Gastrointestinal system surgery patients
* Individuals with pollen allergy

  * Koivuranta PONV risk factors:

Female gender, Non-smoking individuals History of PONV History of motion sickness Anesthesia duration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-01-09 (Actual); Study Completion 2018-02-19 (Actual)

PRIMARY OUTCOMES:
PONV Occurence in all Participants by Rhodes Index of Nausea, Vomiting and Retching(R-INVR) Scores (8 items; each 0-4 points;total of 0-32 points) | Early postoperative period; 0-6 hours after surgery
  PONV measure; Any score above zero (>0) indicates that participant experienced nausea.
  Each response is scored as 0: minimum, 4: maximum disturbance, and the score from 8 items was summed. The worst PONV experience can be expressed with the highest value of 32 points. 3 subscales were "experience, occurence, and distress".
  Experience (total experience score; 32):
  Nausea Experience Questions: 4,5,7; Total score; 0-12 Vomiting Experience Questions: 1,3,6; Total score; 0-12 Retching Experience Questions: 2,8; Total score; 0-8
  Occurence (total occurence score; 20):
  Nausea Occurence Questions: 4,7; Total score; 0-8 Vomiting Occurence Questions: 1, 6; Total score; 0-8 Retching Occurence Questions: 8; Total score; 0-4
  Distress (total occurence score; 12):
  Nausea Distress Questions: 5; Total score; 0-4 Vomiting Distress Questions: 3; Total score; 0-4 Retching Distress Questions: 2; Total score; 0-4
The Comparison of PONV Occurence by total R-INVR Scores in the Intervention and Control Groups | Early postoperative period; 0-6 hours after surgery
  PONV measure; Any R-INVR total score above zero (>0) indicates that participant experienced nausea. This results were compared in control and intervention groups.
The Comparison of PONV Intensity by Total score of R-INVR (0-32 points) in the Intervention and Control Groups | Early postoperative period; 0-6 hours after surgery
  R-INVR scale total score was summed; higher points indicate worse nausea and/or vomiting Each response is scored between 0 to 4, and the score from 8 items were summed. The worst PONV experience can be expressed with the highest value of 32 points. These scores were compared in control and intervention groups and analysed.
The Comparison Between R-INVR Average Scores in the Intervention and Control Groups | Early postoperative period; 0-6 hours after surgery
  R-INVR scale total score was averaged in groups (total score0-32 points by 8 items each 0-4 points) (control, intervention); higher score indicates worse nausea and/or vomiting within the group
The Comparison of R-INVR Average Scores by the Intervention and Control groups | Early postoperative period; 0-6 hours after surgery
  R-INVR scale averaged scores were compared in groups (control, intervention); higher score indicates worse nausea and/or vomiting within the group.
Visual Analog Scale (VAS) (0-10 points) for PONV | Early postoperative period; 0-6 hours after surgery
  The level of experienced nausea and vomiting described by participants and nurses using VAS; 10 indicates the worst experience of nausea and/or vomiting; and 0, no nausea or vomiting being experienced

SECONDARY OUTCOMES:
Anesthesia duration by minutes (marked as sign in and time out) and PONV occurence (R-INVR total score) comparison | Early postoperative period; 0-6 hours after surgery
  Anesthesia duration (by minutes; defined risk factor) was compared with PONV occurence (measured with total R-INVR score)
The Comparison of Smoking status (smoking or not smoking) of Participants in the Intervention and Control Groups was compared with PONV occurence (R-INVR total score) | Early postoperative period; 0-6 hours after surgery
  People who do not smoke (tobacco) is proved to be under risk for PONV and this status was compared with R-INVR total score.
The Comparison of intraoperative Intravenous Ondansetron and PONV occurence (R-INVR total score >0) in All Participants | Early postoperative period; 0-6 hours after surgery
  Ondansetron use (by patient who received (4 or 8 mg IV during surgery, the dose was determined by anesthesia residents depending on patients' weight, verses patients who did not receive any ondansetron at all during surgery) was analysed against PONV occurence (R-INVR total score>0 or 0)
The Comparison of intraoperative Intravenous Ondansetron and PONV occurence (R-INVR total score >0) in All Participants in the Intervention and Control Groups | Early postoperative period; 0-6 hours after surgery
  Ondansetron use (by patient who received (4 or 8 mg IV during surgery, the dose was determined by anesthesia residents depending on patients' weight, verses patients who did not receive any ondansetron at all during surgery) was compared by PONV occurence (R-INVR total score>0 or 0) in control and intervention groups
The Comparison of the Intensity of PONV Occurence in PONV risk groups (not smoking, women, age <50, over one hour anesthesia, previous experience of PONV or motion sickness) by the total R-INVR scores | Early postoperative period; 0-6 hours after surgery
  The intensity of experienced PONV measured by the total score of R-INVR was analysed according to risk factors (not smoking, women, age <50, over one hour anesthesia, previous experience of PONV or motion sickness)
Gender (men or women) and PONV relation | Early postoperative period; 0-6 hours after surgery
  Woman gender is a described risk factor for PONV and R-INVR results by gender were comprised.
Age and PONV relation | Early postoperative period; 0-6 hours after surgery
  Younger age is a described risk factor for PONV and R-INVR results for PONV were analysed for a relation between R-INVR scores with participants' age. A linear relation was analysed if the R-INVR scores declined by age or not.
Age over and below 50 and PONV relation | Early postoperative period; 0-6 hours after surgery
  The participants' data was divided in two according to age by being over or below 50 years; this was a described risk factor and R-INVR total scores were analysed for a relation between PONV and participants' age.

CONTACTS AND LOCATIONS:
Overall Officials: OYA GUMUSKAYA, PhD, Principal Investigator — Yeditepe University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The raw data will be available after consensus reached within investigators regarding publication and following publication of all study results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 2 years from publication of all results.
Access Criteria: Contact to investigators.